CLINICAL TRIAL: NCT00319150
Title: Resistance to ErythroPoietin Effectiveness Algorithm Trial
Brief Title: REPEAT Study - Resistance to ErythroPoietin Effectiveness Algorithm Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: New evidence and trouble recruiting
Sponsor: Queen's University (Other)
Collaborators: Ortho Biotech, Inc. (Industry)
Responsible Party: Dr. Karen E. Yeates, Queens University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMED-852-05
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Kidney Failure, Chronic; Drug Resistance
Keywords: Erythropoetin resistance; End Stage Renal Disease on hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Erythropoietin; Eosinophil Peroxidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (No Intervention): Epo dose to remain constant throughout study
- Dosage Decrease Arm (Active Comparator): Arm 2 is to have an decrease of erythropoietin at regular intervals.
  Interventions: Drug: erythropoietin

INTERVENTIONS:
Drug: erythropoietin — Decrease dosage by 12.5% q 2 weeks according to an algorithm.
  Other Names: Epo
  Arms: Dosage Decrease Arm

SUMMARY:
A strategy for optimizing erythropoietin therapy in patients with erythropoietin resistance. A multi-centered, open-label, randomized, controlled trial.

DETAILED DESCRIPTION:
Study Rationale

Many treatable causes of erythropoietin resistance (also known as erythropoietin hypo-responsiveness) exist in patients with chronic kidney disease (CKD) stages 3 to 5 . Well recognized causes of erythropoietin resistance include iron deficiency, severe hyperparathyroidism, chronic infection, vitamin deficiency, aluminum toxicity and poor dialysis adequacy. Furthermore, many diseases resulting in the chronic inflammatory state have also been associated with erythropoietin resistance in Non-CKD patients with diseases such as chronic congestive heart failure, chronic liver disease and many connective tissue diseases including rheumatoid arthritis and systemic lupus.

It is now well recognized that CKD stage 5 patients receiving dialysis may also be at risk of developing chronic inflammation resulting in a more severe syndrome characterized by malnutrition and resistance to exogenous erythropoietin replacement therapy. Markers of a chronic inflammatory state that are observed in dialysis patients include hypoalbuminemia, elevated C-reactive protein (CRP), elevated ferritin, increased serum amyloid A and low transferrin saturation. In addition, pro-inflammatory cytokines such as interleukin 6 (IL-6), tumour necrosis factor alpha (TNF-alpha) and interleukin 1 (IL-1) have been shown in vivo to suppress erythroid colony forming units. Erythrocyte lifespan can also be shortened through increased clearance by macrophages that are activated by inflammatory signals and immunoglobulin coated erythrocytes.

Inflammation also affects iron metabolism at many levels. Inflammatory cytokines can lead to reduced serum concentrations of iron and transferrin. Reduction in transferrin then leads to decreased iron absorption via the gut. Lactoferrin in polymorphonuclear cells can act as an iron scavenger with bactericidal activity. Lactoferrin levels have been shown to increase in inflammation and can bind large amounts of free iron, thereby reducing overall availability. Functional iron deficiency, which is also a characteristic the inflammatory state associated with erythropoietin resistance is defined as low availability of iron for erythropoiesis despite normal or high iron stores. Functional iron deficiency can occur in two ways; when high doses of exogenous erythropoietin stimulate erythropoiesis and it exceeds the capacity to deliver adequate iron or alternatively, when delivery of iron from the reticuloendothelial system to hematopoietic cells is blocked. Both mechanisms may occur in patients with chronic inflammation and erythropoietin resistance.

Erythropoietin resistance has been defined in several ways. In studies that analyzed Eprex® use, authors have utilized a dose cut off point of >200units of Eprex®/kg/week as a reasonable marker of 'true' erythropoietin resistance, or erythropoietin resistance occurring with no obvious cause contributing to a poor Eprex® response. Other authors have used the dose cut point of >300units /kg/week to define erythropoietin resistance. Furthermore, a measure of erythropoietin resistance called the Eprex® dose to hematocrit ratio (Eprex®/Hct) has been used as a continuous variable in some studies and has been shown to be positively correlated with certain markers of erythropoietin resistance.

Markers of erythropoietin resistance in dialysis patients have been studied. Previous studies have shown that CRP levels greater than 20mg/L are associated with Eprex® resistance in dialysis patients. Other markers include low albumin, high fibrinogen, low transferrin and high ferritin. Other novel markers of inflammation such as plasma N-acetyl-seryl-aspartyl-lysyl-proline, procalcitonin, fetuin and neopterin have also been studied.

The true prevalence of Eprex® resistance is not known in Canada. It is estimated to be approximately 10% based on the early Eprex® therapy trials. The Canadian Nephrology Practice Patterns Study (CNPPS), which collected data on a large subset of Canadian dialysis patients from 1995 to 1998 provides some further estimates. Several authors have analyzed the CNPPS data and applied Eprex® resistance measures to this study population. Using the dose cut off point of >200units/kg/week of Eprex®, the authors found that the prevalence of Eprex® resistance was 15.7% for hemodialysis (HD) patients and 5.5% for peritoneal dialysis (PD) patients. Further analysis using the Eprex®/Hct measure showed a significant negative correlation between Eprex®/Hct and serum albumin in both HD and PD patients. Body mass index (BMI) was also positively correlated with Eprex®/Hct in both groups. This study also found that when the dose cut off of >200units/kg/week was utilized as a measure of exogenous erythropoietin resistance, 15% of the HD patients above this cut off point were utilizing 34% of all the Eprex® administered to HD patients in the study period. Similarly, 5.5% of Eprex® resistant PD patients required 16.2% of all the Eprex® given to PD patients during the same period.

Little is known about the optimal way to manage 'true' erythropoietin resistance or erythropoietin hypo-responsiveness. Traditionally, nephrologists have overcome erythropoietin resistance by prescribing large or escalating Eprex® doses over prolonged periods of time. There is minimal data that suggests the optimal way to manage these patients. There are no published protocols that have studied systematic increases or decreases in Eprex® in such patients. Furthermore, there are few studies on the safety of the use of high dose Eprex® over prolonged periods of time. It is not known whether a dose ceiling beyond which Eprex® is no longer pharmacologically effective exists in patients with 'true' Eprex® resistance. Studies into the cost effectiveness of high dose Eprex® therapy in Eprex® resistant patients are limited.

Patients with Eprex® resistance may be able to maintain their hemoglobin levels on reduced dose Eprex®, but evidence for the efficacy and safety of an Eprex® dose reduction protocol is limited to small open-label studies. In contradistinction, perhaps escalating Eprex® doses to a maximum dose well above the recommended clinical practice guideline target is what is required to improve hemoglobin levels in these patients.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* Adult patients > 18 years old with current Epoetin Alpha dose >250 units/kg/wk
* Hemoglobin >90g/L or <130g/L
* Patients whom a temporary fall in Hb of up to 10g/L is deemed safe
* Patients not expected to have a change in the type of Epo or route of Epo therapy for the duration of the Study period

Exclusion Criteria:

* Known iron deficiency (% saturation <20 or ferritin <100)
* Vit B12 or folate deficiency (levels below normal limit for centre lab)
* Known malignancy (solid organ, leukemia or multiple myeloma)
* Jehovah's witness patients/those who refuse transfusion
* Expected to die in the next 6 months
* On dialysis less than 3 months
* Temporary (not tunneled) dialysis access catheter
* Pure red cell aplasia
* High likelihood of early withdrawal or interruption of the study (eg. severe or unstable coronary artery disease, stroke, severe liver disease within the 12 weeks before screening)
* Planned major elective surgery during the study period
* Pregnancy or breast-feeding
* Women of child-bearing potential without effective contraception (abstinence, oral contraceptives, diaphragm, IUD)
* Administration of another investigational drug within 4 weeks before screening or planned during study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Primary End-points: | December 31, 2009
Eprex® dose at the completion of the study period | December 31, 2009
Hemoglobin at completion of the study period (average of last 2 Hb measurements) | December 31, 2009

SECONDARY OUTCOMES:
Number of transfusions of packed red cells | December 31, 2009
# of active infections during the study period (active infection is defined in Appendix B) | December 31, 2009
Hospitalization | December 31, 2009
Difference in HRQOL scores using Renal SF-36 scores taken at study start and completion study completion | December 31, 2009
Death | December 31, 2009

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Yeates, MD, FRCP(C), MPH, Principal Investigator — Queens University
Locations (7):
- Canada (7):
  - Foothills Hospital, Calgary, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Memorial University Medical Centre, St. John's, Newfoundland and Labrador
  - Kingston General Hospital, Kingston, Ontario
  - London Helath Sciences Centre, London, Ontario
  - Humber River Regional Hosptial, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario